CLINICAL TRIAL: NCT00006418
Title: Molecular Genetics of Schizophrenia
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Other Study IDs: R01MH059571 (NIH); R01MH059571 (NIH); R01MH059588 (NIH); R01MH060870 (NIH); R01MH059565 (NIH); R01MH059566 (NIH); R01MH060879 (NIH); R01MH059586 (NIH); R01MH061675 (NIH); R01MH059587 (NIH); DNBBS 7G-GRR
Record Dates: First submitted 2000-10-25; First posted 2000-10-26 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2005-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Genetics
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Procedure: DNA collection

SUMMARY:
This study will create a DNA collection with blood samples from families with at least two siblings who have schizophrenia symptoms. This collection will help scientists identify genes that predispose people to schizophrenia.

DETAILED DESCRIPTION:
Each site will recruit individuals in a large geographic area, and use efficient ascertainment strategies and assessment procedures in order to maximize the number collected. Subjects thought to have schizophrenia will be assessed by personal and family interviews and a review of medical records. Diagnoses will be made by consensus best-estimate procedures. Blood specimens will be obtained from all individuals with schizophrenia or schizoaffective disorder plus their available parents and also the control individuals. A clinical self-assessment will be administered to each control subject. The assessment will include validated self-assessments of lifetime major depression, anxiety disorders, and substance use, and self-reported history of bipolar or psychotic symptoms. Permanent cell lines will be created and DNA extracted at the NIMH-sponsored Center for Genetic Studies. At the end of the four-year project period, biological materials and blinded pedigree and clinical data will be made available to the scientific community for genetic studies of schizophrenia and related disorders. The control sample will, however, be released in a staggered fashion, twice during each fiscal year, to start during the 2nd year of recruitment. The informed consent for controls includes consent for specimens to be used in research on the genetics of any medical disorder. In years 3 and 4, we will undertake association analyses. Power analyses suggest that this study will have excellent power to detect loci associated with genes with relatively small etiologic effects. Data derived from this study will potentially have applications for the treatment and prevention of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals thought to have schizophrenia or schizoaffective disorder, be the parent of such an individual, or be in the matched control group of unrelated individuals not thought to have schizophrenia or schizoaffective disorder

Exclusion Criteria:

* Unable to give informed consent to all aspects of the study
* Psychotic disorder judged to be secondary to substance use, psychotic disorder that appears to be secondary to a known medical or neurological disorder, or severe mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10800 (Estimated)
Dates: Start 2003-09; Study Completion 2007-08

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - University of California, Irvine, Irvine, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Evanston Northwestern Healthcare Research Institute, Evanston, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
- University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Suarez BK, Duan J, Sanders AR, Hinrichs AL, Jin CH, Hou C, Buccola NG, Hale N, Weilbaecher AN, Nertney DA, Olincy A, Green S, Schaffer AW, Smith CJ, Hannah DE, Rice JP, Cox NJ, Martinez M, Mowry BJ, Amin F, Silverman JM, Black DW, Byerley WF, Crowe RR, Freedman R, Cloninger CR, Levinson DF, Gejman PV. Genomewide linkage scan of 409 European-ancestry and African American families with schizophrenia: suggestive evidence of linkage at 8p23.3-p21.2 and 11p13.1-q14.1 in the combined sample. Am J Hum Genet. 2006 Feb;78(2):315-33. doi: 10.1086/500272. Epub 2006 Jan 3. PMID 16400611
- [Background] GAIN Collaborative Research Group; Manolio TA, Rodriguez LL, Brooks L, Abecasis G; Collaborative Association Study of Psoriasis; Ballinger D, Daly M, Donnelly P, Faraone SV; International Multi-Center ADHD Genetics Project; Frazer K, Gabriel S, Gejman P; Molecular Genetics of Schizophrenia Collaboration; Guttmacher A, Harris EL, Insel T, Kelsoe JR; Bipolar Genome Study; Lander E, McCowin N, Mailman MD, Nabel E, Ostell J, Pugh E, Sherry S, Sullivan PF; Major Depression Stage 1 Genomewide Association in Population-Based Samples Study; Thompson JF, Warram J; Genetics of Kidneys in Diabetes (GoKinD) Study; Wholley D, Milos PM, Collins FS. New models of collaboration in genome-wide association studies: the Genetic Association Information Network. Nat Genet. 2007 Sep;39(9):1045-51. doi: 10.1038/ng2127. PMID 17728769
- [Background] Sanders AR, Duan J, Levinson DF, Shi J, He D, Hou C, Burrell GJ, Rice JP, Nertney DA, Olincy A, Rozic P, Vinogradov S, Buccola NG, Mowry BJ, Freedman R, Amin F, Black DW, Silverman JM, Byerley WF, Crowe RR, Cloninger CR, Martinez M, Gejman PV. No significant association of 14 candidate genes with schizophrenia in a large European ancestry sample: implications for psychiatric genetics. Am J Psychiatry. 2008 Apr;165(4):497-506. doi: 10.1176/appi.ajp.2007.07101573. Epub 2008 Jan 15. PMID 18198266
- [Background] O'Donovan MC, Craddock N, Norton N, Williams H, Peirce T, Moskvina V, Nikolov I, Hamshere M, Carroll L, Georgieva L, Dwyer S, Holmans P, Marchini JL, Spencer CC, Howie B, Leung HT, Hartmann AM, Moller HJ, Morris DW, Shi Y, Feng G, Hoffmann P, Propping P, Vasilescu C, Maier W, Rietschel M, Zammit S, Schumacher J, Quinn EM, Schulze TG, Williams NM, Giegling I, Iwata N, Ikeda M, Darvasi A, Shifman S, He L, Duan J, Sanders AR, Levinson DF, Gejman PV, Cichon S, Nothen MM, Gill M, Corvin A, Rujescu D, Kirov G, Owen MJ, Buccola NG, Mowry BJ, Freedman R, Amin F, Black DW, Silverman JM, Byerley WF, Cloninger CR; Molecular Genetics of Schizophrenia Collaboration. Identification of loci associated with schizophrenia by genome-wide association and follow-up. Nat Genet. 2008 Sep;40(9):1053-5. doi: 10.1038/ng.201. PMID 18677311
- [Background] O'Donovan MC, Norton N, Williams H, Peirce T, Moskvina V, Nikolov I, Hamshere M, Carroll L, Georgieva L, Dwyer S, Holmans P, Marchini JL, Spencer CC, Howie B, Leung HT, Giegling I, Hartmann AM, Moller HJ, Morris DW, Shi Y, Feng G, Hoffmann P, Propping P, Vasilescu C, Maier W, Rietschel M, Zammit S, Schumacher J, Quinn EM, Schulze TG, Iwata N, Ikeda M, Darvasi A, Shifman S, He L, Duan J, Sanders AR, Levinson DF, Adolfsson R, Osby U, Terenius L, Jonsson EG, Cichon S, Nothen MM, Gill M, Corvin AP, Rujescu D, Gejman PV, Kirov G, Craddock N, Williams NM, Owen MJ; Molecular Genetics of Schizophrenia Collaboration. Analysis of 10 independent samples provides evidence for association between schizophrenia and a SNP flanking fibroblast growth factor receptor 2. Mol Psychiatry. 2009 Jan;14(1):30-6. doi: 10.1038/mp.2008.108. Epub 2008 Sep 23. PMID 18813210
- [Background] Psychiatric GWAS Consortium Coordinating Committee; Cichon S, Craddock N, Daly M, Faraone SV, Gejman PV, Kelsoe J, Lehner T, Levinson DF, Moran A, Sklar P, Sullivan PF. Genomewide association studies: history, rationale, and prospects for psychiatric disorders. Am J Psychiatry. 2009 May;166(5):540-56. doi: 10.1176/appi.ajp.2008.08091354. Epub 2009 Apr 1. PMID 19339359
- [Background] Shi J, Levinson DF, Duan J, Sanders AR, Zheng Y, Pe'er I, Dudbridge F, Holmans PA, Whittemore AS, Mowry BJ, Olincy A, Amin F, Cloninger CR, Silverman JM, Buccola NG, Byerley WF, Black DW, Crowe RR, Oksenberg JR, Mirel DB, Kendler KS, Freedman R, Gejman PV. Common variants on chromosome 6p22.1 are associated with schizophrenia. Nature. 2009 Aug 6;460(7256):753-7. doi: 10.1038/nature08192. Epub 2009 Jul 1. PMID 19571809
- [Background] Gejman PV, Sanders AR, Duan J. The role of genetics in the etiology of schizophrenia. Psychiatr Clin North Am. 2010 Mar;33(1):35-66. doi: 10.1016/j.psc.2009.12.003. PMID 20159339
- See also: National Institute of Mental Health Center for Genetic Studies — http://zork.wustl.edu/nimh